CLINICAL TRIAL: NCT05310734
Title: A Single Treatment Pharmacokinetic and Safety Study of Natroba (Spinosad) Topical Suspension 0.9% w/w in Subjects 1 Month to 3 Years 11 Months of Age With an Active Scabies Infestation
Brief Title: PK and Safety Study of Natroba Topical Suspension 0.9% in Subjects 1 Month to 3 Years 11 Months of Age With Scabies
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cipher Pharmaceuticals Inc. (Industry)
Collaborators: Concentrics Research (Other); Iqvia Pty Ltd (Industry); Medpace, Inc. (Industry); Inotiv Laboratories (Unknown); BioAgilytix (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SPN-110-21
Record Dates: First submitted 2022-03-09; First posted 2022-04-05 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-02

CONDITIONS: Scabies
Keywords: Pharmacokinetics; PK; Pharmacokinetics and Safety Study of Spinosad; PK and Safety Study of Spinosad; Spinosad PK and Safety Study; Safety; Pharmacokinetic and Safety Study of Natroba; PK and Safety Study of Natroba; Natroba PK and Safety Study
MeSH Terms: conditions — Scabies | interventions — spinosad; Benzyl Alcohol

STUDY DESIGN:
Intervention Model Description: A blood draw will be taken from subjects just before a full body spinosad application (t=0) and then at 0.5 and 3.0 hours. The following PK parameters will be calculated for spinosad (spinosyn A and spinosyn D) and benzyl alcohol in each subject: Cmax, Tmax, and Area Under the Curve (AUC) 0-3h. Safety assessments include monitoring of AEs, general skin and eye irritation, laboratory assessments, prior medications, and concomitant medications. Smaller laboratory blood samples will be collected pre-dose and 3-hours post-dose prior to discharge.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- PK and Safety (Experimental): A Single 6-hour Treatment, Pharmacokinetic and Safety Study of Natroba (spinosad) Topical Suspension 0.9% w/w in Subjects 1 Month to 3 Years 11 Months of Age with an Active Scabies Infestation.
  Interventions: Drug: Spinosad Topical

INTERVENTIONS:
Drug: Spinosad Topical — A topical suspension indicated for the treatment of scabies is used for this PK and Safety Study
  Other Names: Natroba; benzyl alcohol

SUMMARY:
A population of approximately 50 pediatric subjects will be enrolled to assess the PK of spinosad and benzyl alcohol for 3 hours following a single, full-body topical application (open label) on a single in-clinic visit (Day 1, or Day 2 if screening only on Day 1). There will be approximately 50 subjects ages 1 month to 3 years 11 months of age enrolled with the goal of completing approximately 16 subjects. With assistance from a caregiver, Natroba will be applied over the entire body from the neck down to the toes (including the soles of the feet) and to the hairline, temples, forehead and possibly the scalp (if a scabies infestation is present on the scalp). The open-label Investigational Product (IP) will remain on the skin for at least 6 hours before removing the IP by gentle washing. The subjects will stay in the clinic until the 3-hour procedures are completed. Blood draws will be taken at 0 hours just prior to treatment, and then at 0.5 and 3.0 hours post-treatment. Heel sticks are likely to be the mode of blood collection for children less than 2 years of age. A ±5-minute time window will be allowed for all post-treatment blood samples. Removal of IP can occur by the caregiver at home after it has been on the skin for at least 6 hours before bathing the child. Safety will be assessed with adverse events (AEs), general skin and eye irritation assessments, and pre-dose and pre-discharge laboratory evaluations. Following the sample collections subjects will be released from the clinic and directed to their primary care physician for follow-up. Subjects will be provided scabies medications upon discharge to dispense to family members. These include 5% Permethrin for those in the household that are less than 4 years of age and Natroba for those in the household 4 years of age and older. Subjects who terminate early will not be given these medications to dispense to family members.

DETAILED DESCRIPTION:
A population of approximately 50 pediatric subjects will be enrolled to assess the PK of spinosad and benzyl alcohol for 3 hours following a single, full-body topical application (open label) on a single in-clinic visit (Day 1, or Day 2 if screening only on Day 1). There will be approximately 50 subjects ages 1 month to 3 years 11 months of age enrolled with the goal of completing approximately 16 subjects. With assistance from a caregiver, Natroba will be applied over the entire body from the neck down to the toes (including the soles of the feet) and to the hairline, temples, forehead and possibly the scalp (if a scabies infestation is present on the scalp). The open-label Investigational Product (IP) will remain on the skin for at least 6 hours before removing the IP by gentle washing. The subjects will stay in the clinic until the 3-hour procedures are completed. Blood draws will be taken at 0 hours just prior to treatment, and then at 0.5 and 3.0 hours post-treatment. Heel sticks are likely to be the mode of blood collection for children less than 2 years of age. A ±5-minute time window will be allowed for all post-treatment blood samples. Removal of IP can occur by the caregiver at home after it has been on the skin for at least 6 hours before bathing the child. Safety will be assessed with adverse events (AEs), general skin and eye irritation assessments, and pre-dose and pre-discharge laboratory evaluations. Following the sample collections subjects will be released from the clinic and directed to their primary care physician for follow-up. Subjects will be provided scabies medications upon discharge to dispense to family members. These include 5% Permethrin for those in the household that are less than 4 years of age and Natroba for those in the household 4 years of age and older. Subjects who terminate early will not be given these medications to dispense to family members.

Natroba (spinosad) Topical Suspension, 0.9% w/w applied by a parent/guardian in a single, full-body topical application from the neck down to the toes (including the soles of the feet) and to the hairline, temples, forehead and possibly the scalp (if a scabies infestation is present on the scalp).

A blood draw will be taken from subjects just before spinosad application (t=0) and then at 0.5 and3.0 hours. The following PK parameters will be calculated for spinosad (spinosyn A and spinosyn D) and benzyl alcohol in each subject: Cmax, Tmax, and Area Under the Curve (AUC) 0-12h.

Safety assessments include monitoring of AEs on study Day 1 or Day 2, general skin and eye irritation assessment on Day 1 or Day 2, laboratory assessments on Day 1 or Day 2, prior medications, and concomitant medications on Day 1 (and Day 2, if applicable). Smaller laboratory blood samples will be collected pre-dose and 12-hours post-dose prior to discharge.

Pharmacokinetic (PK) parameters will be calculated by using model independent methods. Standard statistical analyses will be done on these parameters for the purpose of interpretation of the data (Cmax, Tmax and Area Under the Curve (AUC) 0-3h and will be used to assess the absorption over 3 hours post-administration in 50 subjects (1 month - 3 years 11 months). The PK parameter estimates will be computed with noncompartmental methods for each subject. Individual elapsed sampling times (actual time) will be used in the PK analysis and parameters will be computed for each subject. Descriptive summaries of the plasma concentration levels for both spinosad (spinosyn A and spinosyn D) and benzyl alcohol observed at each nominal time point will be provided. Descriptive summaries of the PK parameter estimates will also be completed. Summary statistics for continuous variables will include number of non-missing observations, mean, standard deviation, coefficient of variation (CV%), median, minimum, and maximum, geometric mean and standard error of the geometric mean.

The safety endpoints include the evaluation of adverse events, general skin and eye irritation assessments, clinical laboratory assessments, and use of prior medications and concomitant medications. Additionally, the descriptive changes from baseline (pre-dose) to final assessment (pre-discharge) will be calculated for applicable parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ages 1 month to 3 years and 11 months.
2. Must have active scabies infestation confirmed by clinical signs and symptoms (evidence of burrows or presence of scabies inflammatory/non-inflammatory lesions and pruritus) as well as by burrow ink test (BIT) to demonstrate the presence of burrowing mites.
3. Generally, in good health based on medical history and clinical assessments.
4. Normal-appearing skin in non-infested areas.
5. No history of chronic or recurrent dermatologic disease.
6. Willingness to comply with the study procedures including blood collections and application of study treatment in-clinic.

Exclusion Criteria:

1. Presence of crusted scabies (Norwegian scabies).
2. Allergies or intolerance to ingredients in the Investigational Product.
3. Known renal or hepatic impairment.
4. Treatment with scabicide within the prior 2 weeks.
5. Immunodeficiency (including HIV infection) as reported in Medical History.
6. Signs or symptoms of systemic infection.
7. Administration of systemic therapy for infectious disease within the prior 2 weeks.
8. Receipt of any investigational product within the prior 4 weeks.
9. Medications used for itching or other indication that contain benzyl alcohol or other alcohols within the past 7 days.
10. Over-the-counter cortisone products within the past 7 days.
11. Oral prescription medications and/or antibiotics within the past 7 days.
12. Any other conditions that, at the investigator's discretion, may interfere with the study conduct, or which might confound the interpretation of the study results, or which may put the subject at undue risk.

Ages: 1 Month to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2022-03-04 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Cmax for Spinosyn A | Blood samples collected up to 3 hours post treatment - 0 (pre-treatment), 0.5 and 3.0 hours post-treatment.
  Peak Plasma Concentration of Spinosyn A in Natroba (spinosad) Topical Suspension, 0.9%
Tmax for Spinosyn A | Blood samples collected up to 3 hours post treatment - 0 (pre-treatment), 0.5 and 3.0 hours post-treatment.
  The time after administration of Natroba (spinosad) Topical Suspension, 0.9% when the maximum plasma concentration is reached for Spinosyn A.
Area Under the Curve (AUC) 0-3 for Spinosyn A | Blood samples collected up to 3 hours post treatment - 0 (pre-treatment), 0.5 and 3.0 hours post-treatment.
  Area under the plasma concentration versus time curve Area Under the Curve (AUC) of Spinosyn A in Natroba (spinosad) Topical Suspension, 0.9%.
Cmax for Spinosyn D | Blood samples collected up to 3 hours post treatment - 0 (pre-treatment), 0.5 and 3.0 hours post-treatment.
  Peak Plasma Concentration of Spinosyn D in Natroba (spinosad) Topical Suspension, 0.9%
Tmax for Spinosyn D | Blood samples collected up to 3 hours post treatment - 0 (pre-treatment), 0.5 and 3.0 hours post-treatment.
  The time after administration of Natroba (spinosad) Topical Suspension, 0.9% when the maximum plasma concentration is reached for Spinosyn D.
Area Under the Curve (AUC) 0-3 for Spinosyn D | Blood samples collected up to 3 hours post treatment - 0 (pre-treatment), 0.5 and 3.0 hours post-treatment.
  Area under the plasma concentration versus time curve Area Under the Curve (AUC) of Spinosyn D in Natroba (spinosad) Topical Suspension, 0.9%.
Cmax for Benzyl Alcohol | Blood samples collected up to 3 hours post treatment - 0 (pre-treatment), 0.5 and 3.0 hours post-treatment.
  Peak Plasma Concentration of benzyl alcohol (above Limit of Quantitation (1.0 μg/mL) in Natroba (spinosad) Topical Suspension, 0.9%.
Tmax for Benzyl Alcohol | Blood samples collected up to 3 hours post treatment - 0 (pre-treatment), 0.5 and 3.0 hours post-treatment.
  The time after administration of Natroba (spinosad) Topical Suspension, 0.9% when the maximum plasma concentration is reached for benzyl alcohol.
Area Under the Curve (AUC) 0-3 for Benzyl Alcohol | Blood samples collected up to 3 hours post treatment - 0 (pre-treatment), 0.5 and 3.0 hours post-treatment.
  Area under the plasma concentration versus time curve Area Under the Curve (AUC) of benzyl alcohol in Natroba (spinosad) Topical Suspension, 0.9%.
Treatment Emergent Adverse Events | Through study completion, 3 hours
  Treatment emergent AEs will be coded using MedDRA and summarized by System Organ Class and Preferred Term.
Change in General Skin Irritation | Through study completion, 3 hours
  The skin assessment will include documentation of presence or absence of irritation.
Change in General Eye Irritation | Through study completion, 3 hours
  The eye assessment will include documentation of presence or absence of irritation with a rating scale 0-3. 0 - no irritation, 1 - mild scleral, lid and/or lid injection with conjuctival erythema; 2 - moderate scleral and/or lid injection with conjunctival erythema; 3 - severe scleral and/or lid injection with conjunctival erythema and purulent drainage.

CONTACTS AND LOCATIONS:
Overall Officials: Sharda Angl, Study Director — Cipher Pharmaceuticals Inc.; Julie Aker, MT(ASCP), Study Chair — Concentrics Research; William Miller, MD, Principal Investigator — Concentrics Research
Locations (3):
- United States (3):
  - L&C Professional Medical Research Institute, Miami, Florida
  - Velocity Clinical Research, Lafayette, Louisiana
  - Elixir Research Group, Houston, Texas

IPD SHARING:
Plan to Share IPD: No